CLINICAL TRIAL: NCT02970045
Title: Norris ORIEN Total Cancer Care Protocol: A Lifetime Partnership With Patients
Brief Title: Norris ORIEN Total Cancer Care
Status: Recruiting | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0S-15-12; NCI-2016-00770 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 0S-15-12 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2016-07-29; First posted 2016-11-21 (Estimated); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Cancer Risk; Malignant Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor tissue, bone marrow, blood, saliva, sputum, urine, feces, hair, surface skin
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ancillary-Correlative (biospecimen collection): Patients undergo collection of blood during a regular care visit or not up to 4 times a year. Extra tissue is collected after removal during standard of care surgery and patients may undergo additional tumor sampling (needle passes) at the time of planned diagnostic biopsies. During bone marrow biopsy, the doctor may reposition the needle up to 3 times, and bone marrow for research will not be collected more than 4 times per year. Patients may undergo additional collection of other biological samples such as saliva, sputum, urine, feces, hair, and surface skin swabs for analysis. Patients also receive surveys or questionnaires to collect demographics, medical, family, and nutritional history, cancer predisposing risk factors, quality of life data, and quality of care data.
  Interventions: Procedure: Biospecimen Collection; Procedure: Evaluation of Cancer Risk Factors; Other: Medical Chart Review; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood, tissue, and other biological samples
Procedure: Evaluation of Cancer Risk Factors — Ancillary studies
  Other Names: cancer risk factors evaluation
Other: Medical Chart Review — Review of medical chart
  Other Names: Chart Review
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This research trial collects biological samples and clinical information to create a repository of data from patients with cancer or a predisposition for cancer. Combining genetic information from biological samples and clinical data may lead to more knowledge about why certain cancers respond to treatment and help create more personalized medicine.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish a longitudinal study of clinical and related data from patients with or at risk for cancer.

II. To establish a large biospecimen repository that is linked to clinical and related data.

III. To follow patients through their lifetime though passive or active follow-up.

IV. To use clinical data, tissues, other biological samples and derived molecular data in the Total Cancer Care Protocol (TCCP) repositories to match patients in this TCCP study to future studies.

OUTLINE:

Patients undergo collection of blood during a regular care visit or not up to 4 times a year. Extra tissue is collected after removal during standard of care surgery and patients may undergo additional tumor sampling (needle passes) at the time of planned diagnostic biopsies. During bone marrow biopsy, the doctor may reposition the needle up to 3 times, and bone marrow for research will not be collected more than 4 times per year. Patients may undergo additional collection of other biological samples such as saliva, sputum, urine, feces, hair, and surface skin swabs for analysis. Patients also receive surveys or questionnaires to collect demographics, medical, family, and nutritional history, cancer predisposing risk factors, quality of life data, and quality of care data.

After completion of study, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Limited to those patients who are registered for outpatient or inpatient care at University of Southern California (USC) Norris
* Able to understand and sign the TCCP informed consent, California subject's bill of rights, Health Insurance Portability and Accountability Act (HIPAA), and research authorization form directly or through an authorized representative; the informed consent, subject's bill of rights, HIPAA, and research authorization will be available in both English and Spanish languages

Exclusion Criteria:

* Individuals who are not registered as patients for outpatient or inpatient care at USC Norris
* Individuals who are unable to understand or sign the TCCP informed consent, subject's bill of rights, HIPAA, and research authorization in either English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cancer or predisposition for cancer recruited from University of Southern California/Kenneth Norris, Jr. Comprehensive Cancer Center and Hospital
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2016-05-02 (Actual); Primary Completion 2036-05-02 (Estimated); Study Completion 2037-05-02 (Estimated)

PRIMARY OUTCOMES:
Number of biospecimen collected for a centralized repository that is linked to clinical data | Up to 21 years
  Establish and maintain a unique repository of blood, tissue, other biological samples and their associated data (survey data, medical records data, cancer registry data, and other related data) collected from thousands of patients 18 years of age or older who have cancer or are at risk of developing cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Bodour Salhia, PhD, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States